CLINICAL TRIAL: NCT02138201
Title: Representation of the Bladder Innervation Using Diffusion Tensor Imaging Fiber Tracking With MRI - a Pilot Study
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2013-25
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Injury; Neurogenic Lower Urinary Tract Dysfunction
Keywords: diffusion tensor imaging fiber tracking; magnetic resonance Imaging; spinal cord injury; neurogenic lower urinary tract dysfunction
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control: individuals with normal bladder function
- neurogenic bladder: individuals suffering from neurogenic lower urinary tract dysfunction

SUMMARY:
The exact innervation of the bladder and the changes after a spinal cord injury have been not yet been illustrated.

Diffusion tensor imaging with magnetic resonance imaging is a new technique which can be used to visualize single nerve fibers, and thus represent the neural supply of a region in vivo. There are studies in which both the sacral plexus and the lumbar nerve roots have been represented using diffusion tensor imaging. However, there is no study concerning the innervation of the bladder.

The investigators are therefore using diffusion tensor imaging with magnetic resonance imaging to represent the bladder innervation of individuals with neurogenic lower urinary tract dysfunction and individuals with normal bladder function.

ELIGIBILITY:
Inclusion Criteria:

* neurogenic lower urinary trat dysfunction
* normal bladder function

Exclusion Criteria:

* no signed informed consent
* contraindications for MRI (pace maker, implanted metal, claustrophobia)
* upper or lower urinary tract surgeries
* pregnancy (anamnestic)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals with and without neurogenic lower urinary trat dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
bladder innervation quality | day 0
  bladder innervation is illustrated using diffusion tensor imaging fiber tracking with magnetic resonance imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland